CLINICAL TRIAL: NCT02247856
Title: IN VIVO ASSESSMENT OF RADIOLABELED AEROSOL DURING NONINVASIVE VENTILATION IN STABLE COPD: A RANDOMIZED CROSSOVER CLINICAL TRIAL
Brief Title: COPD AND ASSESSMENT OF RADIOLABELED AEROSOL DURING NONINVASIVE VENTILATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniella Cunha Brandao (Other)
Collaborators: Universidade Federal de Pernambuco (Other)
Responsible Party: Sponsor-Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Valdecir_COPD
Record Dates: First submitted 2014-09-21; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: COPD
Keywords: nebulizers,; noninvasive ventilation; COPD; scintigraphy,; aerosol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Noninvasive ventilation+ jet nebulizer
  Interventions: Other: Noninvasive ventilation; Device: Jet Nebulizer
- Experimental Group (Experimental): Noninvasive ventilation+ Vibrating Mesh Nebulizer (VMN)
  Interventions: Other: Noninvasive ventilation; Device: Vibrating Mesh Nebulizer (VMN)

INTERVENTIONS:
Other: Noninvasive ventilation — Bilevel positive pressure (BiPAP Synchrony, Respironics®, Murrysville, Pennsylvania, USA) was applied through face mask (Comfort Full 2, Respironics®, Murrysville, Pennsylvania, USA) attached with straps and pressure adjusted were 12 cmH2O of inspiratory pressure and 5 cmH2O of expiratory pressure after a period of adaptation before beginning the procedure to avoid ventilator-patient asynchrony
Device: Jet Nebulizer — Both nebulizers were charged with 2.5 mg of salbutamol and 0.25 mg of ipratropium bromide and 3 mL of saline solution was added to complete 3 Ml. JN (Mist yMax, Air Life, Yorba Linda, USA) was positioned in the circuit using a "T" piece, particle size generation in a 5 µm range (according to the manufacturer information) and flow oxygen tritated at 8 L/min
  Arms: Control Group
Device: Vibrating Mesh Nebulizer (VMN) — Both nebulizers were charged with 2.5 mg of salbutamol and 0.25 mg of ipratropium bromide and 3 mL of saline solution was added to complete 3 Ml. VMN (Aeroneb Solo, Galway, Ireland) was positioned in the mask using an elbow (Elbow Kit, Respironics®, Murrysville, Pennsylvania, USA), particle size generation in a 1 µm and connected to electrical energy.
  Arms: Experimental Group

SUMMARY:
Background: Beneficial effects from noninvasive ventilation (NIV) in acute COPD are well-established, but couple to nebulization is still challenging. Aim: To compare radioaerosol pulmonary deposition and radioaerosol mass balance in the different compartments (pulmonary and extrapulmonary) using vibrating mesh nebulizer (VMN) and jet nebulizer (JN) coupled to NIV.Methods: It was a crossover study involving 9 stable moderate to severe COPD randomly allocated for both phases of the study: Phase 1(NIV+MN,n=9) and phase 2(NIV+JN,n=9). Bronchodilators were delivered during NIV using a facemask (pressures of 12 cmH2O and 5 cmH2O - inspiratory and expiratory, respectively). Radioactivity counts were performed using a gamma camera and regions of interest(ROIs) were delimited. We determine aerosol mass balance from the lungs, upper airways, stomach, nebulizer, circuit, inspiratory and expiratory filters, and mask as a percentage.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were considered as follows: moderate to severe stable COPD (50% ≤ FEV1 < 80% from predicted values or 30% ≤ FEV1 < 50% from predicted values)(4); none exacerbation in the last six months; age between 18 - 60 years; both sexes; no smoking history; able to understand verbal commands, and consent to participate in this protocol.

Exclusion Criteria:

Presence of dyspnea; cardiopulmonary diseases (chronic obstructive pulmonary disease, pneumonia, cardiac failure, myocardial infarction, pneumothorax); hyperthermia; hemodynamic instability (heart rate > 150 bpm and systolic blood pressure < 90 mmHg); arrhythmia absence; pregnancy; and contraindications for use of NIV (29).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
radioaerosol deposition index into the lungs | 10 months
  Immediately after inhalation, participants sat in a chair with the back positioned in front to the gamma camera (STARCAM 3200 GE, California, USA) to obtain radioactivity counts from the posterior thorax during a period of 300 seconds on a matrix of 256 X 256. After, participants were positioned sitting in front to the gama camera to obtain images from face. Then, the same procedure was performed to analysis deposition in the nebulizer, circuits, inspiratory filter, expiratory filter and face mask. Counts representing stomach were obtained from posterior thorax and corrections for decay of technetium were used to during extrapulmonary measurements

SECONDARY OUTCOMES:
radioaerosol mass balance that reached pulmonary and extrapulmonary compartments. | 10 months
  The analysis of deposition in pulmonary and extrapulmonary compartments was expressed as a percentage from the count in each compartment to the total radioaerosol mass generated by nebulizers. The inhaled radioaerosol was considered the sum of deposition into the upper airways, lungs and stomach.
  Regions of interest were delimited based on a previous protocol and RDI was expressed as absolute values and was calculated according to the counts generated from each regions of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Valdecir G Filho, PhD, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Hospital das Clínicas de Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Brandao DC, Lima VM, Filho VG, Silva TS, Campos TF, Dean E, de Andrade AD. Reversal of bronchial obstruction with bi-level positive airway pressure and nebulization in patients with acute asthma. J Asthma. 2009 May;46(4):356-61. doi: 10.1080/02770900902718829. PMID 19484669
- [Result] Galindo-Filho VC, Brandao DC, Ferreira Rde C, Menezes MJ, Almeida-Filho P, Parreira VF, Silva TN, Rodrigues-Machado Mda G, Dean E, Dornelas de Andrade A. Noninvasive ventilation coupled with nebulization during asthma crises: a randomized controlled trial. Respir Care. 2013 Feb;58(2):241-9. doi: 10.4187/respcare.01371. PMID 22781558
- [Result] Soroksky A, Stav D, Shpirer I. A pilot prospective, randomized, placebo-controlled trial of bilevel positive airway pressure in acute asthmatic attack. Chest. 2003 Apr;123(4):1018-25. doi: 10.1378/chest.123.4.1018. PMID 12684289